CLINICAL TRIAL: NCT04839926
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase I Clinical Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of CY150112 After Single Oral Administration in Healthy Chinese Subjects
Brief Title: A Single Ascending Dose Study Of CY150112 After Single Oral Administration in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: NH101-11
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia
Keywords: Safety, Tolerability,Pharmacokinetics; CY150112; Single Ascending Dose
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0.5mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 0.5mg CY150112
- 1.5mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 1.5mg CY150112
- 4.5mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 4.5mg CY150112
- 10mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 10mg CY150112
- 18mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 18mg CY150112
- 24mg CY150112 (Experimental): single oral CY150112 while fasting on day 1.
  Interventions: Drug: 24mg CY150112

INTERVENTIONS:
Drug: 0.5mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 0.5mg CY150112
Drug: 1.5mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 1.5mg CY150112
Drug: 4.5mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 4.5mg CY150112
Drug: 10mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 10mg CY150112
Drug: 18mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 18mg CY150112
Drug: 24mg CY150112 — single oral CY150112 while fasting on day 1.
  Other Names: placebo
  Arms: 24mg CY150112

SUMMARY:
The primary objective of single ascending dose study is to evaluate the safety and tolerability of CY150112 after single oral administration of different doses in healthy Chinese subjects.

DETAILED DESCRIPTION:
Single administration, double-blinded, placebo-controlled (2 subjects in each group will take placebo,8 subjects in each group will take CY150112) and 6 dose groups (0.5mg, 1.5mg, 4.5mg, 10mg, 18mg and 24mg).

This study comprises a screening period (between signing of the informed consent form and Day -1), baseline period (Day -1), treatment period (Days 1-5) and follow-up period(Days 12 or 7 days after discharge ).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subjects are 18<age ≤45 years of age when signing the informed consent.
2. Male Subjects with body weight of ≥50.0kg ，and female Subjects with body weight of ≥45.0kg and BMI (body mass index) of 18.5≤ and <28.0 at screening examination.
3. After detailed explanations of study objectives, contents and procedures, and possible risks, subjects are aware of all relevant information related to this study and have signed the written informed consent form voluntarily.
4. Subjects are able to communicate well with researchers, be willing and able to comply with the lifestyle restrictions stipulated during this study period, and cooperate to complete this study.

Exclusion Criteria:

1. The investigator determined that the subjects' present medical history and past medical history had any disease or dysfunction that would affect the clinical trial, including but not limited to diseases of the central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, hematological system, etc.
2. There is any surgical condition or disease that may significantly affect the absorption, distribution, metabolism and excretion of drugs, or may harm to the subjects participating in the trial; such as history of gastrointestinal operations (gastrectomy, gastroenterostomy, enterectomy, etc.), urinary tract obstruction or dysuria, gastroenteritis, digestive tract ulcers, history of gastrointestinal bleeding, etc.
3. Subjects with past history of allergy to drugs or allergic disease.
4. Subjects with currently or past history of mental disorders and brain functional disorders.
5. According to the Columbia suicide severity scale (C-SSRS), subjects were at risk of suicide or were at risk of suicide based on the clinical judgment of the researchers, or with past history of self-injurious behavior.
6. Subjects have history of drug abuse or positive urine drug tests at screening within 1 year prior.
7. Subjects have history of alcohol abuse(i.e.,criteria are per week consumption more than 14 standard units(1 unit =360mL beer or 45mL 40% alcohol of Chinese liquor or 150mL wine)or positive alcohol breath tests at screening within 1 year prior.
8. Average amount of daily smoking>5 cigarettes at screening 3 months prior.
9. Those who have special requirements for food, cannot follow a uniform diet or have difficulty swallowing.
10. Female subjects who are pregnant and lactating ; and those who refuse to use effective non-drug contraceptive measures (such as abstinence, intrauterine device) or have planned to donate sperm or ovum throughout the study period and within 3 months after the end of the study.
11. Abnormal vital signs, lab and ECG indicators, as determined by the researcher, and clinically significant (e.g., male QTC > 450ms female > 470ms,corrected by Friericia ).
12. Subjects who resting heart rate <55 beats/min or >100 beats/min; systolic blood pressure <90mmHg or >140mmHg; diastolic blood pressure <60mmHg or >90mmHg.
13. Subjects who hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab), or HIV antibody (HIV-Ab), or syphilis serum reaction (TRUST) is non-negative.
14. Subjects who glutamic-pyruvic transaminase(ALT), creatinine (Cr), urea nitrogen (BUN) exceeding the normal upper limit or the level of serum prolactin is 2 times higher than the normal upper limit.
15. Subjects who participated in any clinical trial within 3 months before medication.
16. Subjects have history of blood donations of 400 mL within 3 months before enrollment; 200 mL within 1 month before enrollment; or have history of using blood products.
17. Subjects who had a history of surgery within 3 months prior to enrollment, or did not recover from surgery, or had an expected surgical plan during the study period.
18. Subjects who had taken any drugs, including prescription and over-the-counter drugs within 2 weeks prior to enrollment.
19. Subjects who directly related to this clinical trial.
20. Subjects have poor compliance or other problems that the researchers believe that it is not suitable for participating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Incidence of Adverse Events

SECONDARY OUTCOMES:
Cmax | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Maximum (peak) observed drug serum concentration
AUC0-t | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) to the time of the dosing interval
AUC0-∞ | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time
%AUCex | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Extrapolation percentage of AUC0-∞
Tmax | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Time of occurrence of Cmax
T1/2 | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Biological half life correlated with the elimination rate constant (kel) of semi-logarithmic concentration-time curve
Vd | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Apparent volume of distribution
CL | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Clearance
λz | pre-dose（within1hour）,0.25,0.5,1,1.5,2,2.5,3,4,6,8,12,24,48,96hours post-dose
  Elimination rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Hua Fang li, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China